CLINICAL TRIAL: NCT07097415
Title: The Application of Continuous Blood Glucose Monitoring in Optimizing the Management of Early Onset and Late Onset Type 2 Diabetes: an Effectiveness - Implementation Type Ⅱ Hybrid Design Quasi-experimental Pragmatic Trial
Brief Title: The Application of Continuous Blood Glucose Monitoring in Optimizing the Management of Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Feng Sun, associate professor, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00001052-24080
Record Dates: First submitted 2025-07-04; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Continuous Glucose Monitoring; Type 2 Diabetes (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGM Group (Experimental): (1) individualized health education sessions conducted by endocrinology healthcare providers covering CGM concepts, usage methods, advantages, risks, and precautions, along with hands-on device demonstration and provision of written materials and user manuals; (2) development of an integrated CGM data management platform that connects with community healthcare information systems for real-time data transmission, storage, and analysis; (3) establishment of standardized CGM response protocols for healthcare providers, including glucose target setting, dietary and exercise recommendations, personalized medication adjustments based on glucose fluctuations, and management procedures for hypoglycemic and hyperglycemic alerts; and (4) mobile application setup and data transmission configuration for patients.
  Interventions: Device: Continuous blood glucose monitoring assisted blood glucose management
- control group (No Intervention): 1. Blood Glucose Monitoring Method Maintain Traditional Self-Monitoring of Blood Glucose (SMBG): Continue using existing traditional blood glucose monitoring methods throughout the 24-week trial period.
     Monitoring Flexibility:
     No restrictions on the frequency or method of daily home blood glucose measurements; No restrictions on the type of traditional blood glucose monitoring devices used Patients can perform blood glucose monitoring according to personal habits and physician recommendations.
  2. Medical Management Routine Medical Care: The control group's routine medication and treatment are not restricted by the study.
  Treatment Adjustments: During the trial period, patients and physicians can make adjustments at any time based on actual blood glucose control status, including:
  Medication adjustments; Dietary modifications; Exercise modifications Non-Intervention Principle: This study does not intervene in any of the above adjustments but requires detailed recording of all changes.

INTERVENTIONS:
Device: Continuous blood glucose monitoring assisted blood glucose management — (1) individualized health education sessions conducted by endocrinology healthcare providers covering CGM concepts, usage methods, advantages, risks, and precautions, along with hands-on device demonstration and provision of written materials and user manuals; (2) development of an integrated CGM data management platform that connects with community healthcare information systems for real-time data transmission, storage, and analysis; (3) establishment of standardized CGM response protocols for healthcare providers, including glucose target setting, dietary and exercise recommendations, personalized medication adjustments based on glucose fluctuations, and management procedures for hypoglycemic and hyperglycemic alerts; and (4) mobile application setup and data transmission configuration for patients.
  Arms: CGM Group

SUMMARY:
This study investigates the effectiveness and implementation of continuous glucose monitoring (CGM) technology for type 2 diabetes management in Chinese community healthcare settings. Type 2 diabetes represents a significant public health challenge in China, with traditional blood glucose monitoring methods presenting limitations including patient discomfort, incomplete glucose data, and delayed information transmission to healthcare providers. CGM devices offer continuous, real-time glucose monitoring with the potential to improve patient outcomes and healthcare delivery efficiency.

This quasi-experimental pragmatic trial employs an effectiveness-implementation Type II hybrid design, enrolling 800 adults with type 2 diabetes from two community health centers in Yinzhou District, Ningbo. Participants are randomly assigned to either a CGM intervention group or a control group using traditional self-monitoring blood glucose methods. The CGM group receives device training and wears CGM systems for three separate 2-week periods over 24 weeks, while the control group continues standard monitoring practices. The primary outcome is change in glycated hemoglobin (HbA1c) levels, with secondary outcomes including other metabolic markers, patient satisfaction, and quality of life measures. Simultaneously, the study explores implementation factors using the Consolidated Framework for Implementation Research (CFIR) through qualitative interviews with healthcare providers and quantitative surveys with patients. This comprehensive approach aims to provide evidence for CGM effectiveness in Chinese patients while identifying barriers and facilitators for successful implementation in community healthcare settings, ultimately informing strategies for improving diabetes management at the population level.

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥ 18 years old; ② There is a previous diagnosis of T2DM in the electronic medical record system of Qianhu Hospital and Fuming Street Community Health Service Center, and the diagnosis has been made for 1 year or more; ③ Resident with permanent registered residence registration who has filed in the health records of residents in Yinzhou District.

Exclusion Criteria:

* ① Pregnant women; ② Type 1 diabetes, adult latent autoimmune diabetes, special type diabetes (such as post pancreatic surgery, monogenic diabetes); ③ Patients who are currently using or have previously used hormone drugs that may affect blood sugar levels; ④ Patients with severe renal insufficiency (eGFR<30ml/m ^ 2, or undergoing hemodialysis); ⑤ Patients with severe liver dysfunction (ALT or AST greater than 3 times the upper limit of normal); ⑥ Tumor patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
glycosylated hemoglobin | At baseline and 24-week endpoint
  Measurement method: Laboratory blood test analysis. Assessment timing: At baseline and at 24-week endpoint. Procedure: Venous blood samples collected by clinical physicians, processed at hospital laboratory facilities.

SECONDARY OUTCOMES:
Fasting plasma glucose (FPG) | At baseline and 24-week endpoint
  Measurement method: Laboratory blood test analysis. Assessment timing: At baseline and 24-week endpoint.
Healthcare Provider and Participant Awareness and Acceptance of CGM | at weeks 0, 8, 16, and 24 during the 24-week study period
  Measurement method: Custom-designed structured questionnaires. Assessment timing: Baseline, follow-up visits, and endpoint.
  Questionnaires used:
  1. Baseline survey questionnaire
  2. CGM group follow-up questionnaire
  3. Endpoint survey questionnaire
Time in Range (TIR) | Three 2-week CGM wearing periods at weeks 0, 8, and 16
  Time in Range (TIR): percentage of time glucose levels are within target range (3.9-10.0 mmol/L).
  Measurement method: Continuous glucose monitoring data analysis using CGM device (Anytime CT3A system).
  Assessment period: Three 2-week CGM wearing periods at weeks 0, 8, and 16.
Standard Deviation (SD) | Three 2-week CGM wearing periods at weeks 0, 8, and 16
  Measurement method: Continuous glucose monitoring data analysis using CGM device (Anytime CT3A system).
  Assessment period: Three 2-week CGM wearing periods at weeks 0, 8, and 16.
Mean Amplitude of Glycemic Excursion (MAGE) | Three 2-week CGM wearing periods at weeks 0, 8, and 16
  Measurement method: Continuous glucose monitoring data analysis using CGM device (Anytime CT3A system).
  Assessment period: Three 2-week CGM wearing periods at weeks 0, 8, and 16.
Health-Related Quality of Life composite | At baseline and 24-week endpoint
  Measurement tool: EQ-5D-5L questionnaire, including:
  EQ-5D-5L descriptive system (5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression); EQ VAS (visual analogue scale, 0-100 scale). Assessment timing: Baseline and 24-week endpoint.
Treatment Costs | Continuous assessment from baseline through 24-week endpoint
  Cost components:
  Direct medical costs: CGM device costs, glucose monitoring supplies, outpatient visits, laboratory tests, medications; Healthcare resource utilization: frequency of hospital visits, emergency department visits, hypoglycemia-related healthcare contacts; Data collection: Patient self-report, medical records, and healthcare claims data; Assessment timing: Continuous throughout 24-week study period.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Qianhu Hospital, Ningbo, Zhejiang
  - Fuming Street Community Health Service Center, Ningbo

IPD SHARING:
Plan to Share IPD: No